CLINICAL TRIAL: NCT01818973
Title: Preoporative Bevacizumab, Radiation Therapy, and XELOX Chemotherapy for Locally Advanced Nonmetastatic Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Associate Professo, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6901061
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Bevacizumab; capecitabine; oxaliplatin; preoporative IMRT
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Bevacizumab; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Neoadjuvant chemotherapy with XELOX: Xeloda, po, 1000mg/m2/12h daily, day 1 in the afternoon until day 15 in the morning; Oxaliplatin, iv, 130mg/m2, day 1; and Bevacizumab, iv, 7.5 mg/kg, day 1, during the first cycle (each cycle has 3 weeks).
  Followed by chemoradiotherapy, 50 Gy/25 fractions during 5 weeks plus 2 cycles XELOX and Bevacizumab: Xeloda, po, 1000mg/m2/12h daily, day 1 in the afternoon until day 15 in the morning; Oxaliplatin, iv, 100mg/m2, day 1; and Bevacizumab, iv, 7.5 mg/kg, day 1.
  6-7 weeks from the last radiation therapy, Total Mesorectal Excision (TME) surgery will be performed.
  3-4 weeks after operation, 3 cycles XELOX (the same as the neoadjuvant chemotherapy) and 2 cycles Xeloda (po, 1000mg/m2/12h daily, day 1 in the afternoon until day 15 in the morning) will be administered.
  Interventions: Drug: Xeloda; Drug: Oxaliplatin; Drug: Bevacizumab; Radiation: Radiation; Procedure: surgery

INTERVENTIONS:
Drug: Xeloda — po, 1000mg/m2/12h daily, day 1 in the afternoon until day 15 in the morning, 8 cycles
  Other Names: Capecitabine
Drug: Oxaliplatin — iv, 130mg/m2, day 1, 1 cycle during neoadjuvant chemotherapy and 3 cycles in adjuvant chemotherapy 100mg/m2, day 1, 2 cycles during concurrent chemoradiotherapy
Drug: Bevacizumab — iv, 7.5 mg/kg, day 1, 3 cycles during neoadjuvant chemotherapy and concurrent chemoradiotherapy
  Other Names: Avastin
Radiation: Radiation — Intensity-modulated radiation therapy, 50 Gy/25 fractions during 5 weeks
Procedure: surgery — Total Mesorectal Excision (TME)

SUMMARY:
We presumed that the addition of a monoclonal antibody Bevacizumab into radiation therapy and combination chemotherapy could results in improved pathologic tumor regression grade (TRG) in locally advanced nonmetastatic rectal cancer.

DETAILED DESCRIPTION:
Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Giving bevacizumab together with radiation therapy and combination chemotherapy before surgery may achieve promising improvements in pCR rates, we designed this Phase II study in patients with T3/4 or N1/2 loco-regionally advanced rectum cancer, to examine the efficacy and safety of the addition of bevacizumab to a regimen of capecitabine and oxaliplatin in combination with pre-operative radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum.
* T3 or T4 adenocarcinoma or node positive colorectal tumours.
* Appropriate staging investigations of the primary tumour, either endorectal ultrasound or pelvic MRI.
* Male or female aged 18 to 70.
* Have a performance status ECOG of 0 or 1.
* Have a life expectancy greater than 6 months.
* Adequate organ function and coagulation parameters as measured by: WBC > 4000/mm3, PLT > 100000/mm3, Hb > 10g/dL, ALT < 1.5X ULN, AST < 1.5X ULN, bilirubin < 1.5mg/dL Serum creatinine < 1.8mg/dL.
* Patient consent.

Exclusion Criteria:

* Known to have clinical or radiological evidence of distant metastases.
* Evidence of intestinal obstruction (except for those after enterostomy).
* Patients with a past history of colorectal surgery (except for enterostomy), chemtherapy, radiation, biotherapy or targeted therapy.
* Pregnant woman OR women of childbearing potential with a positive pregnancy test at baseline or lactating.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Patients with a past or current history (within last 5 years) of other malignancies, except for the indication under this study and curatively treated basal and squamous skin cancer or in-situ cancer of the cervix.
* Patients with mental disorder unable to complete the informed consent.
* Uncontrolled hypertension.
* Clinically significant (i.e. active) cardiovascular disease for example:

cerebrovascular accidents (<=6 months), myocardial infarction (<= 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.

* Moderate or serious proteinuria.
* Known hypersensitivity against experimental drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-06 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The pathologic tumor regression grade (TRG) | March 30, 2015

SECONDARY OUTCOMES:
5-y overall survival | March 30, 2020
Occurence of toxicity | March 30, 2015
5-y local relapse free survival | March 30, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yu X, Wang QX, Xiao WW, Chang H, Zeng ZF, Lu ZH, Wu XJ, Chen G, Pan ZZ, Wan DS, Ding PR, Gao YH. Neoadjuvant oxaliplatin and capecitabine combined with bevacizumab plus radiotherapy for locally advanced rectal cancer: results of a single-institute phase II study. Cancer Commun (Lond). 2018 May 21;38(1):24. doi: 10.1186/s40880-018-0294-z. PMID 29784042